CLINICAL TRIAL: NCT06369987
Title: Visual Performance of Dailies Total1 Multifocal and Acuvue Oasys Max 1-Day Multifocal in Presbyopic Lens Wearers
Acronym: GIRAFFE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Waterloo (Other)
Collaborators: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 46238
Record Dates: First submitted 2024-04-12; First posted 2024-04-17 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Presbyopia
MeSH Terms: conditions — Presbyopia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Dailies Total1 Multifocal, ACUVUE OASYS MAX 1-Day Multifocal (Experimental): Fit participant with Dailies Total1 Multifocal first, and with ACUVUE OASYS MAX 1-Day Multifocal second.
  Interventions: Device: Deleficon A (multifocal); Device: Senofilcon A (multifocal)
- ACUVUE OASYS MAX 1-Day Multifocal, Dailies Total1 Multifocal (Experimental): Fit participant with ACUVUE OASYS MAX 1-Day Multifocal first, and with Dailies Total1 Multifocal second.
  Interventions: Device: Deleficon A (multifocal); Device: Senofilcon A (multifocal)

INTERVENTIONS:
Device: Deleficon A (multifocal) — Daily disposable silicone hydrogel contact lenses indicated for presbyopia, in addition to myopia or hyperopia.
  Other Names: Dailies Total1 Multifocal
Device: Senofilcon A (multifocal) — Daily disposable silicone hydrogel contact lenses indicated for presbyopia, in addition to myopia or hyperopia
  Other Names: ACUVUE OASYS MAX 1-DAY Multifocal

SUMMARY:
The purpose of this study is to measure the logMAR visual acuity when presbyopic soft lens wearers are fit with Dailies Total1 Multifocal and ACUVUE OASYS MAX 1-DAY Multifocal.

ELIGIBILITY:
Inclusion Criteria:

1. Are at least 42 years of age and has full legal capacity to volunteer;
2. Have signed an information consent letter;
3. Are willing and able to follow instructions and maintain the appointment schedule;
4. Habitually wears soft contact lenses for the past 3 months (minimum);
5. Are presbyopic and require a reading addition of at least +0.75D and no more than +1.75D;
6. Can be refracted and achieve monocular spectacle distance vision of at least 20/25 Snellen (or +0.10logMAR) visual acuity;
7. Have contact lens power requirements that fall within the available study lens parameters (distance sphere: +6D to -9D; near addition as per each lens design);
8. Can be fit with the initial fitting guidelines provided by the lens manufacturer and use either Low or Medium Add (same add in both eyes).

Exclusion Criteria:

1. Are a current habitual wearer of Dailies Total1 Multifocal or ACUVUE OASYS MAX 1-DAY Multifocal;
2. Has refractive astigmatism higher than -0.75DC in either eye;
3. Are participating in any concurrent clinical or research study involving intervention or invasive ocular tests;
4. Have any known active ocular disease and/or infection;
5. Has a systemic condition that in the opinion of the investigator may affect a study outcome variable;
6. Are using any systemic or topical medications that in the opinion of the investigator may affect a study outcome variable;
7. Have known sensitivity to the diagnostic pharmaceuticals to be used in the study;
8. Have undergone refractive error surgery;
9. Are a member of the Centre for Ocular Research & Education (CORE) directly involved in the study.

Min Age: 42 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2024-04-25 (Actual); Primary Completion 2024-11-21 (Actual); Study Completion 2024-11-21 (Actual)

PRIMARY OUTCOMES:
High contrast visual acuity (logMAR) at 6m | Day 1
  High contrast visual acuity (logMAR) for the dominant eye under photopic illumination at 6m
High contrast visual acuity (logMAR) at 40cm | Day 1
  High contrast visual acuity (logMAR) for the dominant eye under photopic illumination at 40cm

CONTACTS AND LOCATIONS:
Overall Officials: Lyndon Jones, PhD, FCOptom, Principal Investigator — Centre for Ocular Research & Education (CORE)
Locations (1):
- Centre for Ocular Research & Education (CORE), Waterloo, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No